CLINICAL TRIAL: NCT04460768
Title: A Multicountry, Multicenter, Retrospective Study Evaluating the Patient Characteristics, Disease Burden, Treatment Patterns, and Patient Journey of Advanced Epithelial Ovarian Cancer Patients: A Korean, Taiwanese, and Australian Secondary Database Study
Brief Title: An INternational Frontline Ovarian Cancer Real World Management Study
Acronym: INFORM
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00028
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
The current study aims to analyze the existing secondary databases from Korea (Sungkyunkwan University, Samsung Medical Center, Seoul), Taiwan (National Taiwan University, Chang-Gung Medical Foundation Linkou Branch and Mackay Memorial Hospital), and Australia (Australian Ovarian Cancer Study [AOCS]) to leverage the already available data in the real-world setting to review the current standard of care in advanced epithelial ovarian cancer cases. The collected data will help provide the required information for assessing the unmet treatment needs in this patient group. The data will also provide the needed information to support any reimbursement activity needed for future novel therapies in this patient group

DETAILED DESCRIPTION:
Ovarian cancer is the eighth most commonly diagnosed cancer (295,414 cases reported in 2018) and the seventh leading cause of cancer-associated mortality (184,799 deaths reported in 2018) in women, worldwide. The increasing trends in the burden of ovarian cancer, coupled with other challenges, such as lack of awareness of ovarian cancer risk factors, lack of adequate screening tools, lack of access to diagnostics, and lack of trained clinicians, contribute to delays in diagnosis, resulting in a high proportion of patients presenting with advanced-stage ovarian cancer associated with high mortality. Over 75% of women with ovarian cancer have been reported to be diagnosed at a late stage with high relapse rates, despite first-line therapy. Studies in Asia have highlighted that about 65%-70% of women with ovarian cancer are diagnosed at an advanced stage. Further, the five-year net survival rate of advanced-stage ovarian cancer in Asia has been found to range from 14% to 41%.

Among the various ovarian cancer subtypes based on histology, epithelial ovarian cancer is the most common type, reported in about 90% of cases. Specifically, type II epithelial ovarian cancer (that includes serous carcinoma, mixed epithelial and stromal carcinoma, undifferentiated carcinomas, and other epithelial carcinoma) accounts for about 66%-73%, 56%, 73%, and 73% in the US, Asia, Europe, and Oceania, respectively. The corresponding rates for type I epithelial ovarian tumors (that include endometrioid, clear cell, mucinous, squamous, and transitional cell carcinomas) have been noted to be 19%-21%, 32.5%, 20.5%, and 20%, respectively. Regarding prognosis, the five-year net survival rate of type II epithelial ovarian cancer that includes serous carcinoma has been found to be low when compared to other subtypes across all regions. Of note, type II epithelial ovarian tumors have been reported to be highly aggressive and usually present at an advanced stage, with poor survival rates. The recurrence or relapse rates have also been noted to be high with epithelial serous ovarian cancer. Furthermore, a strong association has been noted between family history of ovarian cancer, a very strong risk factor, and the risk of developing aggressive serous carcinomas. Genetic (both germline and somatic) mutations in BRCA1/2 have been noted in about 22% of high-grade, serous, ovarian carcinomas, and the majority of hereditary cases (~44%). Also, mutations in homologous recombination response genes have been noted in about 50% of high-grade serous epithelial ovarian cancer cases.

Considering the high incidence, poor prognosis, and high morbidity and mortality from advanced epithelial ovarian cancer, it is important to have well-organized databases on the clinical characteristics, treatment patterns, and outcomes of these patients, to help identify the unmet needs and gaps and further optimize the survival outcomes in these patients. With exception of the UK, France, Germany, Italy, and Spain and the USA, there is paucity of databases, registries, or published literature on patient level data pertaining to treatment patterns, clinical characteristics, and outcomes of advanced ovarian cancer patients. Therefore, the current study aims to analyze the existing secondary databases from Korea (Sungkyunkwan University, Samsung Medical Center, Seoul), Taiwan (National Taiwan University, Chang-Gung Medical Foundation Linkou Branch and Mackay Memorial Hospital), and Australia (Australian Ovarian Cancer Study) to leverage the already available data in the real-world setting to review the current standard of care in advanced epithelial ovarian cancer cases. The collected data will help provide the required information for assessing the unmet treatment needs in this patient group. The data will also provide the needed information to support any reimbursement activity needed for future novel therapies in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects above the age of 18
* Patients with a confirmed diagnosis of advanced-stage (FIGO III/IV) epithelial (Serous [high or low grade], mucinous, endometrioid, clear cell, mixed, and others) ovarian cancer between the period Jan 2014 and Dec 2018, provided at least 12 months data is available (not mandatory to be ovarian cancer related) as a proxy of healthcare use prior to the diagnosis of advanced-stage epithelial ovarian cancer

Exclusion Criteria:

* Patients being included in interventional clinical trials with PARPi for the treatment of advanced-stage high-grade epithelial ovarian cancer treatment during the study period
* Patients with early stage disease (FIGO Stage I, IIA, IIB, or IIC)
* Other malignancies within the past five years, except adequately treated non-melanoma skin cancer; curatively treated in situ cancer of the cervix; ductal carcinoma in situ; stage 1, grade 1 endometrial carcinoma; or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localized breast cancer may have been eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and remained free of recurrent or metastatic disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a non-interventional study that involves retrospective collection of data from medical records of all patients who have been newly diagnosed with advanced-stage epithelial ovarian cancer (high grade serous type epithelial ovarian cancer for Taiwan) between the period Jan 2014-Dec 2018.
Sampling Method: Probability Sample
Enrollment: 989 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  In first line setting - length of time from diagnosis to first progression, death, or last follow-up. In second line setting, length of time from start of second line therapy until patient has disease progression, death, or last follow-up.

SECONDARY OUTCOMES:
Platinum free interval | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  The number of months elapsed from the last day of platinum chemotherapy for first line of treatment to the date of diagnosis of disease recurrence or date of last follow-up if the patient did not recur during the study period
Time to progression | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  The length of time from the date of cancer diagnosis or the start of anti-cancer treatment until the cancer starts to get worse or spread to other parts of the body.
Duration of treatment | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  The length of time from the start of anti-cancer treatment to end of anti-cancer treatment
Time to first subsequent treatment | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  The length of time from the date of cancer diagnosis to the start of cancer treatment after cancer progression
Overall survival | Retrospective study of patients diagnosed between the period Jan 2014-Dec 2018
  Duration from the index date to the date of death (if available)

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site, Melbourne, Victoria, Australia
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, New Taipei City
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- See also: D0817R00028_CSR_v1.0_clean_0823 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00028&attachmentIdentifier=30b554f7-0338-4254-9a8f-a528fc2c1e33&fileName=D0817R00028_CSR_v1.0_clean_0823_r_Redacted.pdf&versionIdentifier=